CLINICAL TRIAL: NCT05787587
Title: A Study of PARG Inhibitor IDE161 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: IDEAYA Biosciences (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDE161-001; KEYNOTE-F86 (Other: Merck Sharp & Dohme LLC); MK-3475-F86 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-03-17; First posted 2023-03-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced or Metastatic Solid Tumors; Breast Cancer; Ovarian Cancer; Prostate Cancer; Endometrial Cancer; Colorectal Cancer; Head and Neck Cancers; Extensive Stage Small Cell Lung Cancer (ES-SCLC); NSCLC
Keywords: PARPi; PARP inhibitor; BRCA; HRD gene alteration; Breast; Ovarian; Advanced solid tumors; Metastatic solid tumors; BRCA 1; BRCA 2; Homologous recombination; PARG; PARG Inhibition; ATM; BARD1; BRIP1; CDK12; CHEK1; CHEK2; FANCL; PALB2; PPP2R2A; RAD51C; RAD51D; RAD54L; NBN; FANCA; HRD+; Endometrial; Pembro; Pembrolizumab; HR genes; genomic instability score; GIS; GI+; gLOH; genomic loss of heterozygosity; MSS; MSI; MMR; PD-L1; ES-SCLC; SCLC; Extensive Stage Small Cell Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Endometrial Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Mental Retardation, X-Linked, With Or Without Seizures, Arx-Related | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Sequential
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Module 1 Part 1: Monotherapy Dose Escalation (Experimental): Participants will be assigned to a dose level.
  Interventions: Drug: IDE-161
- Module 1 Part 2: Monotherapy Dose Expansion (Experimental): After a dose is decided in Part 1, participants entering part 2 will be assigned to a dose level.
  Interventions: Drug: IDE-161
- Module 2 Part 1: Combination Dose Escalation with pembrolizumab (Experimental): Participants will be assigned to a dose level.
  Interventions: Drug: IDE-161; Drug: Pembrolizumab
- Module 2 Part 2: Combination Dose Expansion with pembrolizumab (Experimental): After a dose is decided in Part 1, participants entering part 2 will be assigned to a dose level.
  Interventions: Drug: IDE-161; Drug: Pembrolizumab

INTERVENTIONS:
Drug: IDE-161 — Oral Medication
Drug: Pembrolizumab — Intravenous Infusion
  Other Names: KEYTRUDA®
  Arms: Module 2 Part 1: Combination Dose Escalation with pembrolizumab; Module 2 Part 2: Combination Dose Expansion with pembrolizumab

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, and efficacy of IDE161 as a single agent and in combination with pembrolizumab.

DETAILED DESCRIPTION:
The purpose of this study is to characterize the safety, tolerability including determination of maximum tolerated dose (MTD), maximum accepted dose (MAD), recommended dose(s) for expansion (RDE) and/or recommended Phase 2 dose (RP2D), pharmacokinetics (PK), pharmacodynamics (PD) and preliminary anti-tumor activity of IDE161 as a single agent in participants with advanced or metastatic solid tumors harboring BRCA1/2 loss of function alterations and/or other defects in the homologous recombination (HR) pathway and in combination with pembrolizumab in participants with advanced/recurrent endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants must be 18 years of age or older
2. Advanced or metastatic solid tumors excluding primary central nervous system (CNS) tumors
3. For Module 1 only, Have documented evidence of BRCA1/2 and/or genetic alterations conferring homologous recombination deficiency (HRD) (ATM, BARD1, BRIP1, CDK12, CHEK1, CHEK2, FANCL, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D, RAD54L, NBN, FANCA)

   For Module 2 only, results of MSI and/or MMR testing required.

   For Module 2 only, results of BRCA1/2 and HRD gene testing required.
4. Participant must have progressed on at least one prior line of therapy in the advanced or metastatic setting that is considered an appropriate standard of care, or for which the participant has documented intolerance
5. For Module 2 only, advanced or metastatic Endometrial Cancer (uterine carcinosarcoma is excluded)
6. For Module 2 only, Must have progressed on treatment with an anti-PD-1/L1 monoclonal antibody (MAB)

Exclusion Criteria:

1. Known primary CNS malignancy
2. Impairment of GI function or GI disease that may significantly alter the absorption of IDE161
3. Have active, uncontrolled infection
4. Clinically significant cardiac abnormalities
5. Major surgery within 4 weeks prior to enrollment
6. Radiation therapy within 2 weeks prior to enrollment
7. Systemic cytotoxic chemotherapy within 4 weeks prior to enrollment
8. Radioimmunotherapy within 6 weeks of enrollment
9. Treatment with a therapeutic antibody within 4 weeks prior to enrollment
10. Treatment with an anti-cancer small molecule within 5 half-lives (t1/2), or 2 weeks, whichever is shorter
11. Have current active liver or biliary disease
12. For Module 2 only, History or allogeneic tissue/solid organ transplant
13. For Module 2 only, Active autoimmune disease that has required systemic treatment in past 2 years
14. For Module 2 only, History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Part 1 (Dose Escalation): To characterize the safety and tolerability of IDE161 monotherapy or in combination with pembrolizumab to determine the MTD and/or RDE | Approximately 2 years
  * Incidence of Dose Limiting Toxicities
  * Incidence of treatment-emergent Adverse Events as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study therapy
  * Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing
Part 2 (Dose Expansion): To further assess the safety and tolerability of IDE monotherapy and in combination with pembrolizumab at the RDE | Approximately 4 years
  * Incidence of treatment-emergent AEs as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study therapy
  * Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE v5.0), and timing
Part 2 (Dose Expansion): To evaluate preliminary anti-tumor activity of IDE161 monotherapy or in combination with pembrolizumab | Approximately 4 years
  Tumor response: Overall Response Rate assessed using RECIST criteria v1.1

SECONDARY OUTCOMES:
Part 2 (Dose Expansion) Assess the risk/benefit at an IDE161 monotherapy dose and exposure alternative to the initial expansion dose; as well as an IDE161 dose in combination with a fixed dose of pembrolizumab and exposure alternative to the initial | Approximately 4 years
  Descriptively compare the totality of emerging data (efficacy, safety, PK, PD) between the initial expansion dose cohort and dose optimization cohort
To characterize the single dose PK Peak Plasma Concentration (Cmax) of IDE161 monotherapy and in combination with pembrolizumab. | Approximately 4 years
  Single-dose PK parameters of IDE161
To characterize the multiple dose PK Peak Plasma Concentration (Cmax) of IDE161 monotherapy and in combination with pembrolizumab. | Approximately 4 years
  Multiple-dose PK parameters of IDE161
To characterize the single dose PK Area under the plasma concentration versus time curve (AUC) of IDE161 monotherapy and in combination with pembrolizumab. | Approximately 4 years
  Single-dose PK parameters of IDE161
To characterize the multiple dose PK Area under the plasma concentration versus time curve (AUC) of IDE161 monotherapy and in combination with pembrolizumab. | Approximately 4 years
  Multiple-dose PK parameters of IDE161
To characterize the single dose PK Time to Peak drug Concentration (Tmax) of IDE161 monotherapy and in combination with pembrolizumab. | Approximately 4 years
  Single-dose PK parameters of IDE161
To characterize the multiple dose PK Time to Peak drug Concentration (Tmax) of IDE161 monotherapy and in combination with pembrolizumab. | Approximately 4 years
  Multiple-dose PK parameters of IDE161

CONTACTS AND LOCATIONS:
Overall Officials: Darrin Beaupre, MD,PhD, Study Director — IDEAYA Biosciences
Locations (27):
- United States (27):
  - HonorHealth Research Institute, Phoenix, Arizona
  - The Angeles Clinic, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - California Pacific Medical Center, San Francisco, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Orlando Health, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - OSF St Francis Medical Center, Peoria, Illinois
  - Indiana University, Indianapolis, Indiana
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Weil Cornell University, New York, New York
  - Sarah Cannon Research Institute - Oklahoma University, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - NEXT Oncology, Irving, Texas
  - NEXT Oncology, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - NEXT Oncology, Fairfax, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin